CLINICAL TRIAL: NCT04180332
Title: Anti Oxidant Enzymes and Total Antioxidant Levels in Diabetes Mellitus Type II Patients and Healthy Individuals With Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajman University (Other)
Responsible Party: Principal Investigator, sudhir rama varma, Assistant Professor, Ajman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NU/CEC/Ph.D04/2010
Record Dates: First submitted 2019-11-23; First posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Periodontal Diseases; Diabetes Mellitus; Enzyme Disorder
Keywords: superoxide dismutase; catalase; anti-oxidant; diabetes mellitus; type 2; periodontitis
MeSH Terms: conditions — Periodontal Diseases; Diabetes Mellitus; Periodontitis | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: cross sectional study
Masking Description: None were masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy (Experimental): The patients were healthy subjects without Periodontal disease or any systemic manifestation
  Interventions: Diagnostic Test: Blood sample
- Periodontal disease without diabetes (Experimental): Patients with periodontal diseases without diabetes
  Interventions: Diagnostic Test: Blood sample
- Periodontal disease with diabetes (Experimental): Patients with periodontal disease and diabetes
  Interventions: Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Blood sample — 5ml of venous blood was taken from the ante cubital vein from each of the study subjects

SUMMARY:
To evaluate the role of antioxidants - superoxide dismutase, catalase, glutathione and total anti oxidant levels in the serum of chronic periodontitis patients and chronic periodontitis with DM Type II patients, then to compare it with healthy controls, to assess their possible role as biomarkers for chronic periodontitis and the possible systemic effects of periodontitis.

DETAILED DESCRIPTION:
This was a cross sectional study involving 300 subjects ,30-60 years of age. 80% was calculated as the power of the study and error was set at 5%. The ethical clearance for the study was obtained from the University central ethics committee. A consent form, was given to all the subjects, which was explained to them and a written consent was taken before enrolling them. As per the prepared case history format, case history was taken for all the subjects who were part of the study The body mass index (BMI) was assessed and subjects who were overweight & obese, with a BMI above 25 , were not included in the study.7 Of the total of 300 subjects,100 subjects who did not have any systemic diseases were included in group I and III, and 100 subjects with diabetes mellitus type II, who were not suffering from any other systemic diseases were included in group II. The diabetic patients in group II were on oral medication (Metformin derivatives) and appropriate diet control measures, for a period of at least one year but not more than five years.

Group I and II patients had chronic generalized severe periodontitis.8 Subjects in group III were systemically healthy and not suffering from any periodontal disease. A single trained investigator examined the periodontal status of all the subjects. Any other type of periodontitis was not included in the study.

Subjects were excluded if they had taken antibiotics any time in the last 4 weeks. Vitamin and mineral supplement intake and those who underwent periodontal treatment procedures in the course of the last 6 months were eliminated from the study. Tobacco users, alcoholics, pregnant as well as lactating women were not included in the study.

Only subjects who had a a RBS score of less than 120 and HbA1c score of less than 7 were accepted in the study.

Then a periodontal examination was carried out, the status of the periodontal condition was determined, and the subjects were alloted to the three groups by the single trained investigator,patient was also referred to a physician to determine the systemic condition.

Following this the patients were allotted to the various groups as per the inclusion criteria. Patients not fulfilling the various criteria were excluded from the study.

5ml of venous blood was taken from the ante cubital vein from each of the study subjects. The blood from each of the subjects was centrifuged and then stored at -20°C. The serum samples were then analysed for the various anti oxidants.

Statistical Analysis Statistical analysis of the data was done using SPSS version 17 software. The comparison of the means of the 2 groups was done using the students 'T' test. Analysis of variance (ANOVA) two tailed test was used to compare the means of more than 2 groups. HSD tukey test with ANOVA jointly,was used to find means that were significantly different from one another. 'p' value (level of significance) less than 0.05 was taken to be statistically significant.

Biochemical Study:

5 ml venous blood which was taken from each study subject was divided into 2 parts. 2 ml of it was collected in EDTA coated vacutainer tubes and 2 ml in plain tubes. The blood in the EDTA coated tubes was used to assess GSH & SOD. The blood in the plain tubes was used to assess the CAT and total antioxidant levels . It was centrifuged and the serum obtained was stored at - 200C for subsequent analysis Superoxide dismutase, glutathione and catalase were assessed by u.v double beam spectrophotometer and total anti-oxidant levels by spectrophotometer.

Total antioxidant capacity of serum was determined by the phosphomolybdenum method . The estimation of superoxide dismutase enzyme was carried out by Beauchamp and Frodovich method. The catalase activity was assessed using the Hydrogen Peroxide reduction method and estimation of glutathione was by the DTNB method.

ELIGIBILITY:
Inclusion Criteria:

* 100 subjects with chronic periodontitis who did not have any systemic diseases were included in group I
* 100 subjects with chronic periodontitis and diabetes mellitus type II, who were not suffering from any other systemic diseases were included in group II, The diabetic patients in group II were on oral medication (Metformin derivatives) and appropriate diet control measures, for a period of at least one year but not more than five years.
* 100 subjects systemically healthy and not having any periodontal disease were included in group III.

Exclusion Criteria:

* Subjects were excluded if they had taken antibiotics any time in the last 4 weeks, or taken vitamin and mineral supplements or underwent periodontal treatment procedures in the course of the last 6 months.
* Tobacco users, alcoholics, pregnant as well as lactating women were also excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Catalase estimation | From baseline to 5 months
  The estimation will be carried out using ELISA biochemical assay

SECONDARY OUTCOMES:
Antioxidant estimation | From baseline to 5 months
  To assess anti-oxidant kevels using ELISA assay

CONTACTS AND LOCATIONS:
Locations (1):
- AB shetty institute of dental sciences, Mangaluru, India

IPD SHARING:
Plan to Share IPD: No